CLINICAL TRIAL: NCT05448781
Title: a Clinical Trial Phase II Prospective, Single-arm Study of Recombinant Human Angioendostatin /PD-1 Mab Combined With First-line Chemotherapy in the Treatment of Driver Gene Negative Advanced Non-small Cell Lung Cancer
Brief Title: Recombinant Human Angioendostatin /PD-1 Mab Combined With First-line Chemotherapy in the Treatment of Driver Gene Negative Advanced NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Endostatin0630
Record Dates: First submitted 2022-07-04; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-06

CONDITIONS: Non Small Cell Lung Cancer; Endostatin
Keywords: NSCLC; endostatin; PD-1 antibody
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Endostatins; Pemetrexed; Paclitaxel; Carboplatin

STUDY DESIGN:
Intervention Model Description: endostatin combined with PD-1 antibody and platinum-containing two-drug chemotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- endostatin combined with PD-1 antibody and platinum-containing two-drug chemotherapy (Experimental): Recombinant human vascular endostatin (Endu): 210 mg (14 PCS), administered by continuous intravenous pumping for 72h every three weeks on the first day of each cycle.Pemetrexed: 500mg/m2, administered intravenously every three weeks on the first day of each cycle.Paclitaxel:175mg/ m2, administered intravenously every three weeks on the first day of each cycle.Albumin paclitaxel:260mg/ m2, administered intravenously every three weeks on the first day of each cycle.
  Carboplatin:5/AUC, maximum dose limited to 600mg, or 75 mg/m2 cisplatin, is administered intravenously every three weeks on the first day of each cycle Tirelizumab: a recommended dose of 200mg/ time, administered every three weeks on the first day of each cycle until disease progression or unacceptable toxicity is developed.
  Interventions: Drug: Endostatin

INTERVENTIONS:
Drug: Endostatin — Eligible patients with advanced NSCLC were treated with endostatin combined with Tirelizumab and platinum-containing two-drug chemotherapy.26 cases of non-squamous cell carcinoma were treated with endostatin combined with Tirelizumab and Pemetrexed+Carboplatin. and 12 cases of squamous cell carcinoma were treated with endostatin combined with Tirelizumab and Paclitaxel/Albumin paclitaxel+Carboplatin,The maintenance treatment phase was continuous treatment with Endu combined with Tirelizumab
  Other Names: Pemetrexed; Paclitaxel; Albumin paclitaxel; Carboplatin; Tirelizumab

SUMMARY:
To evaluate the efficacy and safety of recombinant human endostatin /PD-1 mab combined with first-line chemotherapy in the treatment of driver gene negative advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
This study is planned to enroll 38 eligible patients in China. Patients who fulfill all the inclusion criteria and none of the exclusion criteria will receive 4-6 cycles of endostatin combined with PD-1 antibody and platinum-containing two-drug chemotherapy.The efficacy of first-line treatment was evaluated every 6 weeks (2 cycles, 42 days). Patients with disease control (CR+ PR+SD) and tolerable adverse reactions were treated for 4-6 cycles,The maintenance treatment phase was continuous treatment with Endu combined with PD-1 antibody, and the efficacy was evaluated every 9 weeks until the end of the study when the investigator considered that the patient was not suitable for continued medication or the efficacy evaluation was disease progression (PD). No other antitumor therapy can be performed during the treatment period. Follow-up of survival was once every 3 months.

ELIGIBILITY:
Inclusion Criteria: Only those who meet all the following inclusion criteria can be enrolled in this study:

1) Patients voluntarily participate in this study and sign informed consent; 2) 18-75 years old, male and female; 3) Advanced or metastatic (stage IIIB, IIIC or IV) NSCLC confirmed by histology or cytology, and no mutation was detected in the driver gene; 4) According to the efficacy evaluation criteria for solid tumor (RECIST1.1), at least one measurable lesion should be used as the target, and the measurable lesion should not have received local treatment such as radiotherapy; 5) ECOG PS of the Eastern tumor cooperative group was 0 ~ 1; 6) Expected survival ≥3 months 7) Patients who have not previously received systematic antitumor therapy, including radiotherapy and chemotherapy, targeted and immunotherapy, or patients who relapsed after postoperative adjuvant chemotherapy followed up for more than 6 months; 8) Major organ functions within 7 days before treatment meet the following criteria:

1. Blood routine examination standards (no blood transfusion within 14 days) : ① Hemoglobin (HB) ≥90g/L; ② Absolute value of neutrophil (ANC) ≥1.5×109/L; ③ Platelet (PLT) ≥80×109/L.
2. Biochemical tests should meet the following standards: ① Total bilirubin (TBIL) ≤1.5 times the upper limit of normal value (ULN); ② Alanine aminotransferase (ALT) and aspartate aminotransferase AST≤2.5ULN, ALT and AST≤5ULN in patients with liver metastasis; ③ serum creatinine (Cr) ≤1.5ULN or creatinine clearance (CCr)≥60ml/min; ④ Serum albumin ≥35g/L.

(4) Doppler ultrasound assessment: Left ventricular ejection fraction (LVEF)≥ normal lower limit (50%).

9) Tissue samples should be provided for biomarker (such as PD-L1) analysis, and newly obtained tissues should be selected. For patients unable to provide newly obtained tissues, 5-8 paraffin sections of 3-5μm thick tissue can be provided for archival preservation up to 2 years before enrollment;

Exclusion Criteria:

* Patients with any of the following conditions will not be enrolled in this study:

  1. Severe allergic reaction to humanized antibodies or fusion proteins;
  2. known hypersensitivity to Endu or any component contained in antibody preparations;
  3. Subjects have been diagnosed as immunodeficient or are receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy within 14 days prior to the study's initial administration and are permitted to use physiological doses of glucocorticoids (≤10mg/ day of prednisone or equivalent);
  4. Subjects with active, known or suspected autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, and hypothyroidism, including but not limited to these diseases or syndromes) were excluded. Subjects with type 1 diabetes, hypothyroidism that requires only hormone replacement therapy, skin conditions that do not require systemic treatment (e.g: vitiligo, psoriasis, or hair loss), or conditions that are not expected to recur in the absence of an external trigger can be enrolled;
  5. Patients with pre-existing serious heart disease, including congestive heart failure, uncontrolled high-risk arrhythmia, unstable angina pectoris, myocardial infarction, and severe valvular disease;
  6. Patients who have previously received targeted drug therapy with vascular endothelial growth inhibitors, such as bevacizumab, sunitinib, sorafenib, imatinib, famitinib, rigafenib, apatinib, anlotinib, etc.
  7. Systemic antitumor therapy, including cytotoxic therapy, signal transduction inhibitors, or immunotherapy (or mitomycin C in the 6 weeks prior to receiving the study drug), was planned within 4 weeks prior to the group or during the duration of the study. Field expanding radiotherapy (EF-RT) was performed within 4 weeks prior to grouping or field limiting radiotherapy was performed within 2 weeks prior to grouping.
  8. Presence of active hepatitis B (HBV DNA ≥ 2000IU/ml or 104copies/ml), hepatitis C (positive hepatitis C antibody, and HCV-RNA higher than the lower limit of analysis).
  9. According to chest X-ray examination, sputum examination and clinical examination, active tuberculosis (TB) infection was determined. Patients with a history of active tuberculosis infection within the previous year, even if treated, should be excluded; Patients with a history of active tuberculosis infection more than one year ago should also be excluded unless the duration and type of antituberculosis therapy previously used are demonstrated to be appropriate.
  10. Patients with BMS with symptoms or symptom control for less than 2 months;
  11. Received major surgical treatment, open biopsy or obvious traumatic injury within 28 days before grouping;
  12. Patients whose imaging shows that the tumor has invaded important blood vessels or the investigator judges that the tumor is highly likely to invade important blood vessels and cause fatal massive bleeding during the follow-up study;
  13. Patients with any evidence or history of bleeding, regardless of severity; Patients with any bleeding or bleeding event ≥CTCAE grade 3 within 4 weeks prior to grouping had unhealed wounds, ulcers or fractures;
  14. Experienced arteriovenous/venous thrombosis events within 6 months, such as cerebrovascular accident (including temporary ischemic attack), deep vein thrombosis and pulmonary embolism;
  15. Concomitant diseases that, according to the investigator's judgment, seriously endanger the patient's safety or affect the patient's ability to complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-07-20 (Estimated); Primary Completion 2023-07-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 1 year
  The time from the first date of first-line treatment until the date of objective disease progression or death.

SECONDARY OUTCOMES:
objective response rate (ORR) | 1 year
  Objective response rate after the given treatment in patients accoeding to the evaluation criteria of RECIST1.1
Overall Survival (OS) | 1 year
  The time from the start of first-line treatment to the date of death due to any cause or the date of last contact (censored observation) at the date of data cut-off.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No